CLINICAL TRIAL: NCT04875702
Title: Treat-to-Target Serum Urate Versus Treat-to-Avoid Symptoms in Gout: A Randomized Controlled Trial
Brief Title: Treat-to-Target Serum Urate Versus Treat-to-Avoid Symptoms in Gout
Acronym: TRUST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Hyon Choi, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P000517; 1U01AR080985-01A1 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol; Naproxen; Colchicine; Solar Activity; Prednisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TTT-SU (Active Comparator): The participants randomized to the Treat-to-Target-Serum Urate (TTT-SU) group will be counseled about gout, generalized lifestyle and dietary issues and will be provided with a three-month supply of allopurinol as well as a treatment to prophylax against attacks that might occur during the up-titration of urate lowering therapy. Allopurinol dose increases will occur until SU concentrations achieve a target level < 6.0 mg/dL.
  Interventions: Drug: Allopurinol; Drug: Naproxen 250 MG; Drug: Colchicine 0.6 mg
- TTASx (Active Comparator): Subjects randomized to the treat-to-avoid-symptoms (TTASx) group will receive the same education as the TTT-SU group. In addition, they will receive anti-inflammatory treatments (naproxen, colchicine, and/or prednisone); enough to treat up to six flares over the ensuing three months.
  Interventions: Drug: Allopurinol; Drug: Naproxen 250 MG; Drug: Colchicine 1.2 mg; Drug: Naproxen 500 Mg; Drug: Prednisone 40 mg

INTERVENTIONS:
Drug: Allopurinol — For the TTT-SU group: The dose titration algorithm for allopurinol increases every 4 weeks by 100 mg until the target serum urate of 6 mg/dL is reached or a patient requires 800 mg per day of allopurinol. Subjects will require a blood draw for SU every 4 weeks until reaching the target.
  For the TTASx group: Subjects randomized to the TTASx group will receive anti-inflammatory treatments (naproxen, colchicine, and/or prednisone) for up to six flares over the ensuing three months. Urate lowering therapy (ULT) will only be offered after the third flare during the trial.
  Other Names: Aloprim, Zyloprim
Drug: Naproxen 250 MG — Naproxen 250 mg p.o. twice daily
  Other Names: Prophylaxis
Drug: Colchicine 0.6 mg — Colchicine 0.6 mg p.o. once daily
  Other Names: Prophylaxis
  Arms: TTT-SU
Drug: Colchicine 1.2 mg — Dose escalation to 0.6 mg p.o. twice daily for patients experiencing breakthrough flares or a dose decrease (0.6 mg p.o. every other day) for patients experiencing gastrointestinal intolerance.
  Other Names: Flare
  Arms: TTASx
Drug: Naproxen 500 Mg — dose escalation to 500 mg twice daily for patients experiencing breakthrough flares.
  Other Names: Flare
  Arms: TTASx
Drug: Prednisone 40 mg — For flare glucocorticoids: prednisone taper for 8 days, starting with 40mg (oral) daily.
  Other Names: Flare
  Arms: TTASx

SUMMARY:
The TRUST study is a randomized, controlled multicenter study to evaluate the management of gout by comparing two commonly used treatment strategies for gout (TTT vs TTASx) to determine the most beneficial for a patient-centered gout outcomes, as well as relevant cardiovascular-metabolic-renal endpoints.

DETAILED DESCRIPTION:
This trial aims to answer a fundamental question in the management of gout by comparing two commonly used treatment strategies for gout (TTT vs TTASx) to determine which is most beneficial for a range of patient-centered gout outcomes, as well as relevant CV-metabolic-renal endpoints.

Designing a scientifically valid and pragmatic clinical trial involves numerous tradeoffs in study design, subject eligibility criteria, and outcome measurement. We have come together as primary care physicians and rheumatologists to consider several alternative designs. We first considered the target study population. Since most rheumatologists believe that the TTT approach is superior, it would be difficult to recruit from rheumatology practices. Thus, we aimed to design a trial that would be feasible to conduct in primary care practices, with an intervention that could primarily be run by nurses and physician assistants. This design would be pragmatic and generalizable to primary care practices outside of the setting of a randomized controlled trial. The trial also needs to incorporate the perspectives of rheumatologists, primary care clinicians, allied specialists, and patients when deciding the key issues to be addressed and how best to answer these questions.76 We convened a modified Delphi Panel (mDP) to solicit input using a formal process of voting and discussion. The Delphi Panel is a commonly used approach in health care for areas where there is less than perfect data to make decisions. It also has been used in the social sciences as a method for formalizing input from multiple parties, using voting and discussion.77,78 We selected a broadly representative group of mDP panelists from four categories of constituents who could inform the trial design: patients, nurses, primary care physicians, and rheumatologists. Two voting rounds were held, including a video conference meeting to discuss all the voting questions and re-vote on items where no consensus had been reached on the first round.

ELIGIBILITY:
To be eligible to be enrolled in the study, each patient must:

1. Provide signed written or electronic informed consent.
2. Be between 18 and 90 years old.
3. Be in a participating primary care practice with at least one visit in the previous 36 months.
4. Be diagnosed with gout by the 2015 ACR/EULAR criteria, with 8 or more points on the 2015 ACR/EULAR criteria scoring algorithm.
5. Have experienced at least one gout flare attributed in the previous 12 months.
6. Have a baseline inter-critical serum urate (SU) ≥ 6.0 mg/dL (at screening or in the 30 days before screening)
7. Be able to swallow pills.
8. Agree to practice effective measures of birth control if of reproductive potential.

Exclusion Criteria

Candidates who meet any of the following criteria will be excluded from the study:

1. Diagnosis of CKD Stage 3B or worse (eGFR < 45 mL/min/ 1.73 m2) at screening
2. More than one subcutaneous tophus on clinical examination at screening
3. Two or more episodes of renal colic in the past 5 years
4. Unable to provide informed consent.
5. AST/ALT > 3 × upper limit of normal (ULN) (within 6 months of entry).
6. Pregnancy, planning pregnancy, or breastfeeding.
7. Patients who have been treated with thiopurines (mercaptopurine (PURINETHOL®), azathioprine (IMURAN®), or thioguanine) in the past 12 months or currently being treated with thiopurines are not eligible for the study. Usage of the thiopurines (azathioprine and mercaptopurine) with allopurinol has been shown to cause a significant drug-drug interaction.
8. Unlikely to survive 2 years because of comorbidities.
9. Currently taking > 200 mg of allopurinol per day or any dose of febuxostat. Patients taking 200 mg or less of allopurinol daily may participate, provided they meet the eligibility criteria for flares and current SU, and they have not had a dose escalation in their allopurinol in the previous 6 months.
10. Patients with known allergic or hypersensitive reactions to allopurinol and not willing to initiate febuxostat if urate lowering is indicated.
11. Subjects that test positive for HLA-B*5801 allele, a genetic marker for severe cutaneous adverse reactions caused by allopurinol and are unwilling to initiate febuxostat if urate lowering is indicated by the study. Subjects of higher risk, including Black/African American, Asian (except Japanese), native Hawaiian, or Pacific Islander descent will be tested at screening.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of gout flare | baseline to two years of follow up
  number of gout flares occurring during two years of follow-up between the TTT-SU and TTASx groups

SECONDARY OUTCOMES:
Quality of life assessment | baseline to two years of follow up
  The Short Form 36 Health Survey Questionnaire (SF-36) questionnaire will be used to assess the health status of study participants by surveying 36 questions in 8 domains of health. A higher score indicates a better health status. For the TRUST study a total physical (score of 10 to 30), functional (a score of 4 to 8) and pain (a score of 2 to 11) will be used as the secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hyon K Choi, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - The University of Alabama at Birmingham, South Birmingham, Alabama
  - UCLA Health, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Boston Medical Center (BMC), Boston, Massachusetts
  - NYU Langone, New York, New York
  - West Virginia University (Including Mobile Clinical Trials Unit), Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No